CLINICAL TRIAL: NCT02421146
Title: The Effect of Transcranial Direct Current Stimulation on Human Brains: A Neuroimaging Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Miklos Argyelan, MD, MD, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 14-623
Record Dates: First submitted 2015-04-13; First posted 2015-04-20 (Estimated); Results first posted 2018-04-30 (Actual); Last update posted 2018-04-30 (Actual); Status verified 2018-03

CONDITIONS: Chronic Schizophrenia
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sham tDCS - Healthy Controls (Sham Comparator): The sham group session will contain 20 minute sessions of transcranial direct current stimulatio , but only the first minute will be with 2mA, then unbeknownst to the subject, the unblinded research assistant will turn off the stimulation.
  Interventions: Device: Transcranial direct current stimulation - Sham
- tDCS - Healthy Controls (Active Comparator): will receive real transcranial direct current stimulation. Real tDCS stimulation will involve ten 20 minute stimulations daily (at 2 mA anode over the left DLPFC while cathode over the right suborbital region) on 5 weekdays of two consecutive weeks
  Interventions: Device: Transcranial direct current stimulation
- Sham tDCS - Patients (Sham Comparator): The sham group session will contain 20 minute sessions of transcranial direct current stimulation as well, but only the first minute will be with 2mA, then unbeknownst to the subject, the unblinded research assistant will turn off the stimulation.
  Interventions: Device: Transcranial direct current stimulation - Sham
- tDCS - Patients (Active Comparator): will receive real transcranial direct current stimulation . Real tDCS stimulation will involve ten 20 minute stimulations daily (at 2 mA anode over the left DLPFC while cathode over the right suborbital region) on 5 weekdays of two consecutive weeks
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — Transcranial direct current stimulation (tDCS) is a form of neurostimulation which uses constant, low current (at 2 mA) delivered to the brain area of interest(anode over the left DLPFC while cathode over the right suborbital region) via electrodes on the scalp.
  Other Names: tDCS
  Arms: tDCS - Healthy Controls; tDCS - Patients
Device: Transcranial direct current stimulation - Sham — Transcranial direct current stimulation (tDCS) is a form of neurostimulation which uses constant, low current (at 2 mA) delivered to the brain area of interest(anode over the left DLPFC while cathode over the right suborbital region) via electrodes on the scalp.
  Other Names: tDCS
  Arms: Sham tDCS - Healthy Controls; Sham tDCS - Patients

SUMMARY:
The purpose of this project is to examine brain function before, during, and after the administration of tDCS (Transcranial Direct Current Stimulation). The brain can perform its job well or poorly depending on many things. The investigators will be using computer tasks and paper and pencil questionnaires to measure the relationship between brain performance and the administration of tDCS. In addition, the study team will be using functional magnetic resonance imaging (fMRI) and related imaging techniques to see how your brain works and compare it with the results we collected from the paper and pencil questionnaires. This study will enroll both schizophrenia patients as well as healthy volunteers without any major psychiatric disorder or physical illness.

DETAILED DESCRIPTION:
This is a placebo condition controlled double blind randomized prospective study where the study team plan to acquire clinical, neurocognitive and imaging data in schizophrenia patients and healthy controls. Those who are eligible for the study will be consented, and will be randomized into either group A or B. The length of the study is four weeks. Subjects in both groups will undergo the same procedure, except that while subjects from group A unbeknownst to them will receive only a sham stimulation of tDCS (placebo condition), the subjects from group B will receive real tDCS stimulation. Real tDCS stimulation will involve ten 20 minute stimulations daily (at 2 mA anode over the left DLPFC while cathode over the right suborbital region) on 5 weekdays of two consecutive weeks, while sham will contain 20 minute sessions as well, but only the first minute will be with 2mA, then unbeknownst to the subject, the unblinded research assistant will turn off the stimulation. The subjects will be told that they can be given either a sham or real stimulation and will be asked at the end of the experiment to fill out a visual analog scale indicating their guess about being in the real or sham arm. Following the first two weeks of the study, there will be a follow up period of two weeks when no stimulation or sham will be administered. Subjects, raters, clinicians and most of the research persons will all be kept blind in regards to their placebo or stimulation status until the end of the study. Research persons analyzing neuroimgaing data will break blindness after subject leaves the study, to continuously monitor neuroimaging findings.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 and 60 years of age
2. Subject is competent to provide informed consent

   Additional inclusion criteria for schizophrenia group:
3. Pt diagnosed with schizophrenia according to DSM V criteria.

Exclusion Criteria:

1. MRI contraindications
2. Person with any kind of neurostimulator or pacemaker, or built in electrical device even if it is MRI safe
3. Skin lesions at the site of electrodes and any documented head or neck dermatological disorder
4. Pregnancy
5. Any major neurological (seizures, sclerosis multiplex, etc) disorder
6. Individuals who are illiterate and/or visually impaired
7. Subjects with history of mental retardation, learning disorders or traumatic brain injury

   Additional exclusion criteria for healthy group:
8. Past or current history of any psychotic illness in the subject or in first degree family members
9. Self report of illicit drug use (except marijuana) in the past. Use of marijuana during the last 3 month.
10. Any use of any psychotropic medications (antipsychotics, SSRI, mood stabilizers, benzodiazepines, stimulants) in the last month.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-04; Primary Completion 2016-09-12 (Actual); Study Completion 2016-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miklos Argyelan, MD, Principal Investigator — The Zucker Hillside Hospital
Locations (1):
- Zucker Hillside Hospital, Glen Oaks, New York, United States

IPD SHARING:
Plan to Share IPD: No
via email request

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sham tDCS - Healthy Controls | tDCS - Healthy Controls | Sham tDCS - Patients | tDCS - Patients
Started | 2 | 4 | 3 | 3
Completed | 2 | 4 | 3 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham tDCS - Healthy Controls | tDCS - Healthy Controls | Sham tDCS - Patients | tDCS - Patients | Total
Number analyzed (Participants) | 2 | 4 | 3 | 3 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 4 | 3 | 3 | 12
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 31 [26 to 36] | 29.5 [25 to 36] | 40.7 [31 to 51] | 38.3 [31 to 45] | 34.8 [25 to 51]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2 | 1 | 5
  Male | 2 | 2 | 1 | 2 | 7
Region of Enrollment [Number; unit: participants]
  United States | 2 | 4 | 3 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: Cognition on the RBANS (Repeatable Battery for the Assessment of Neuropsychological Status) Scale
Description: Standard neuropsychological assessment taking approximately 30 minutes. We report here the total score ndifference between 12th day and baseline. Scores at 12th day and at baseline are calculated according to the RBANS standards as following: five index scores are computed from the RBANS (immediate memory, language, visuospatial, attention, delayed memory) that are combined to provide the Total Score. The Total Score is expressed as a standardized score normalized to a population mean of 100, with a standard deviation of 15 (possible scores 40-135). Higher scores reflect better performance. For the detailed procedures and ranges please see: Randolph C, Tierney MC, Mohr E, Chase TN (June 1998). "The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS): preliminary clinical validity". J Clin Exp Neuropsychol. 20 (3): 310-9. doi:10.1076/jcen.20.3.310.823. PMID 9845158. It is a simple delta score: calculating the difference between 12th day and baseline.
Time Frame: baseline (0th day), 12th day
Population: We calculated differences in the cognitive measure (RBANS TScore) before and after tDCS treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham tDCS - Healthy Controls | tDCS - Healthy Controls | Sham tDCS - Patients | tDCS - Patients
Number analyzed (Participants) | 2 | 4 | 3 | 3
units on a scale | 7 (8.49) | 5.25 (17.84) | -1.5 (4.95) | -1.33 (4.73)

2. Secondary Outcome: Cognition on the RBANS ( Repeatable Battery for the Assessment of Neuropsychological Status) Scale. Change Between 26th Day and Baseline.
Description: Standard neuropsychological assessment taking approximately 30 minutes. We report here the total score ndifference between 26th day and baseline. Scores at 26th day and at baseline are calculated according to the RBANS standards as the following: five index scores are computed from the RBANS (immediate memory, language, visuospatial, attention, delayed memory) that are combined to provide the Total Score. The Total Score is expressed as a standardized score normalized to a population mean of 100, with a standard deviation of 15 (possible scores 40-135). Higher scores reflect better performance. For the detailed procedures and ranges please see: Randolph C, Tierney MC, Mohr E, Chase TN (June 1998). "The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS): preliminary clinical validity". J Clin Exp Neuropsychol. 20 (3): 310-9. doi:10.1076/jcen.20.3.310.823. PMID 9845158. It is a simple delta score: calculating the difference between 26th day and baseline.
Time Frame: baseline (0th day), 26th day
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham tDCS - Healthy Controls | tDCS - Healthy Controls | Sham tDCS - Patients | tDCS - Patients
Number analyzed (Participants) | 2 | 4 | 3 | 3
units on a scale | 0.5 (7.8) | -7 (11.5) | -9.5 (6.4) | -0.7 (5.7)

ADVERSE EVENTS:
Arm/Group | Sham tDCS - Healthy Controls | tDCS - Healthy Controls | Sham tDCS - Patients | tDCS - Patients
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/4 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/2 | 0/4 | 0/3 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No